CLINICAL TRIAL: NCT04166162
Title: Businesses That Care - Zacatecas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: AB InBev Foundation (Unknown)
Responsible Party: Principal Investigator, Eric Brown, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20190141
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Alcohol Drinking
Keywords: Underage Drinking
MeSH Terms: conditions — Alcohol Drinking; Underage Drinking | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Focus Group (Experimental): The Focus Group consists of the participating parents who are BTC employees with child/children in the range of 8 to 16 years old. The Focus Group will receive a total of 6 weekly sessions of the TBD Intervention.
  Interventions: Behavioral: Tomando Buenas Decisiones (TBD) Intervention
- Social Development Strategy (SDS) Group (Experimental): All participating BTC workers will be receiving SDS intervention for a minimum of 1 session.
  Interventions: Behavioral: Social Development Strategy (SDS) Intervention
- Brief Intervention Motivational Interviewing (BIMI) Group (Experimental): Participating 11 to 16 year old children of BTC employees will be receiving the BIMI intervention.
  Interventions: Behavioral: Brief Intervention Motivational Interviewing (BIMI) Intervention
- Business that Care (BTC) Coalition Group (Experimental): Participating BTC employees who are selected by the respective directors of the participating companies to be part of the BTC Coalition will receive a total of 8 BTC training sessions in the space of 6 months.
  Interventions: Behavioral: BTC Training Session

INTERVENTIONS:
Behavioral: Brief Intervention Motivational Interviewing (BIMI) Intervention — BIMI is a 15-minute brief interview in person or via video chat with participating youth. The interview will be focused on discussing the impact of drinking alcohol on one's health and how to set personal goals so that alcohol use does not become a problem. A follow up phone or video call at 3 and 6 months post initial interview will also be conducted which will track on the progress of setting and keeping personal goals.
  Arms: Brief Intervention Motivational Interviewing (BIMI) Group
Behavioral: Tomando Buenas Decisiones (TBD) Intervention — The program is adapted from the Guiding Good Choices (GGC) program and will be conducted by a trained facilitator lasting for about 2 hours per session. The program discusses about the best ways to help one's child make good decisions with regards to avoiding alcohol, drugs, and other problem behaviors that may not be healthy to them as well as ways to have good communication and good connections within one's family.
  Arms: Focus Group
Behavioral: Social Development Strategy (SDS) Intervention — SDS is a 2 hour broad-focused environmental intervention consisting of short presentations and workshops designed to provide skills and models for positive human interaction between employees to fellow employees, employees to their children and employees to their supervisors.
  Arms: Social Development Strategy (SDS) Group
Behavioral: BTC Training Session — BTC training session consists of trainings, discussions and tools focused on community mobilization for the assessment and implementation of evidence-informed preventive interventions addressing community health and behavior problems. Each training session lasts about 4 hours.
  Arms: Business that Care (BTC) Coalition Group

SUMMARY:
The purpose of this study is to develop and implement a community-based prevention initiative to prevent youth alcohol use and abuse in Zacatecas, Mexico.

ELIGIBILITY:
Inclusion Criteria for Parent Participants:

* Must be 18 years or older who are actively working at one of the four BTC participating companies in Zacatecas, Mexico.
* Must be residents of the Cities of Zacatecas or Guadalupe, in the state of Zacatecas, Mexico.
* Workers who are illiterate or otherwise literary challenged are included.
* Must have at least one child (biological, step or adopted) between the ages of 8 and 16 years of age.

Exclusion Criteria for Parent Participants:

* Doesn't speak Spanish.

Inclusion Criteria for Children Participants:

* Must be a child (biological, step or adopted) of a BTC employee who participated in the study.
* Must be between the age of 11 to 16 years.

Exclusion Criteria for Children Participants:

* Doesn't speak Spanish.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Sustainability of BTC coalition | 1 year
  Sustainability of the BTC coalition is assessed via the number of coalition members that continues the implementation of the BTC prevention program one year after BTC training.
Change in risk behaviors in TBD Intervention Recipients | Baseline, 6 weeks
  The efficacy of the TBD intervention is assessed via the changes in targeted risk and protective measures on the pre and post TBD survey. Risk factor measures with multiple items is scored by taking the average of all items in the scale. Lower scores are indicative of less risk and of positive effects of the intervention. The average scores are: minimum =1 and maximum = 4.
Change in risk behaviors in SDS Intervention Recipients | Pre-SDS Intervention, Post-SDS Intervention (2 hours)
  The efficacy of the SDS intervention is assessed via the SDS survey. The SDS survey is coded and scored by taking the average of all items in the scale. The higher scores are indicative of greater use of the SDS as an intervention strategy. The average scores are: minimum =1 and maximum = 4.
Change in risk behaviors in BIMI Intervention Recipients | Baseline, 6 months
  The efficacy of the BIMI intervention is assessed via the Care, Relax, Alone, Forget, Friends, Trouble (CRAFFT) survey. The CRAFFT survey consist of 8 questions answered with "yes" or "no". Each No response is scored 0 and each Yes response is scored 1. The total score ranges from 0-8 with the lower score indicating increased positive response to BIMI intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Brown, Principal Investigator — University of Miami
Locations (1):
- Business That Care Participating Companies, Zacatecas City, Mexico

IPD SHARING:
Plan to Share IPD: No